CLINICAL TRIAL: NCT00149851
Title: A Study to Assess the Efficacy, Safety and Tolerability of Tegaserod Alone and in Combination With Omeprazole Given Orally in Patients With Symptoms of Symptomatic Gastroesophageal Reflux Disease (sGERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919B2203
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2008-01

CONDITIONS: Symptomatic Gastroespohageal Reflux Disease
Keywords: GERD, heartburn, regurgitation, reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Gastroesophageal Reflux Disease (GERD) is a common disorder caused by the reflux of gastric (stomach) acid into the esophagus. The exposure of the lining of the esophagus to the acid will cause damage to the esophagus over time. The symptoms of GERD include heartburn and acid regurgitation This study will determine if Tegaserod alone and in combination with omeprazole is safe and relieves the symptoms of heartburn.

ELIGIBILITY:
Inclusion Criteria:

* History of physician diagnosed GERD
* Heartburn and Regurgitation 3 Days during the week prior to screening

Exclusion Criteria:

* History of erosive esophagitis, Barrett's esophagus, esophageal stricture, scleroderma, Zollinger-Ellison Syndrome, known primary disorder
* History or presence of infection or inflammation of the small or large intestine, gastrointestinal malignancy, history of upper GI surgery
* Use of PPI during the last four weeks prior to screening

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 832
Dates: Start 2004-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing resolution of heart-burn during week 4 of treatment
Proportion of patients experiencing resolution of heart-burn during week 4 of treatment in combination with Omeprazole and compared with Omeprazole alone
Decreasing frequency of regurgitation during week 4 of treatment
Decreasing frequency of regurgitation during week 4 of treatment in combination with Omeprazole and compared with Omeprazole alone

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Novartis, East Hanover, New Jersey, United States